CLINICAL TRIAL: NCT05325645
Title: A Multicenter, Placebo-controlled, Randomized, Double-blind, Parallel-group Comparison Trial to Investigate the Efficacy and Safety of Brexpiprazole Once-weekly (QW) Formulation in Patients With Acute Schizophrenia
Brief Title: Trial of Brexpiprazole Once-weekly (QW) Formulation in Patients With Acute Schizophrenia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Collaborators: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 331-102-00062
Record Dates: First submitted 2022-04-06; First posted 2022-04-13 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Acute Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Brexpiprazole QW 48mg (Experimental): Brexpiprazole QW 48mg, tablet, once weekly, for seven weeks(Initial dose Brexpiprazole QW 24mg)
  Interventions: Drug: OPC-34712FUM/ Brexpiprazole fumarate
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OPC-34712FUM/ Brexpiprazole fumarate — 2 brexpiprazole QW tablets 24 mg (48 mg/dose) will be orally administered once weekly for 7weeks.(As an initial dose, one brexpiprazole QW tablet 24 mg and one placebo tablet will be orally administered (24 mg/dose))
  Arms: Brexpiprazole QW 48mg
Drug: Placebo — Two placebo tablets will be orally administered once weekly for 7weeks.
  Arms: Placebo

SUMMARY:
Confirm the efficacy of the brexpiprazole QW formulation versus placebo for acute symptoms of schizophrenia

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years of age and below the age of 65 at the time of informed consent
* Patients with a diagnosis of schizophrenia based on DSM-5® (295.90) (multiple episodes, currently in acute episode) and confirmed by the Mini International Neuropsychiatric Interview (M.I.N.I.) at the time of informed consent
* Patients who are hospitalized, or judged to require hospitalization, for acute relapse of schizophrenia at the time of informed consent
* Patients whose current episode developed within 2 months prior to screening
* Patients who were treated with antipsychotics at appropriate doses for appropriate durations for the most recent acute episode and who are considered to have responded to the antipsychotics (excluding clozapine)
* Patients who experienced a recurrence or exacerbation of symptoms during an antipsychotic-free period
* Patients who have been fully informed of and understand the objectives, procedures, risks, and expected medicinal benefits of the trial and are able to provide written informed consent prior to initiation of any trial-related procedures

Exclusion Criteria:

<Regarding indication>

* Patients presenting a first episode of schizophrenia based on the clinical judgment of the investigator
* Patients who are considered resistant/refractory to antipsychotic treatment Patients who are "unresponsive to medication with 2 or more antipsychotics at effective doses for a sufficiently long duration (6 weeks)" will be deemed resistant/refractory to antipsychotic treatment.
* Patients who have a history of treatment with clozapine for schizophrenia
* Patients experiencing acute depressive symptoms within 30 days prior to informed consent that, in the judgment of the investigator, require treatment with an antidepressant
* Patients who fall under any of the following criteria regarding suicidal ideation and suicidal behavior

  * Patients who answered "yes" to Question 4 "Active Suicidal Ideation with Some Intent to Act, without Specific Plan" or Question 5 "Active Suicidal Ideation with Specific Plan and Intent" regarding C-SSRS suicidal ideation at screening (for the past 6 months) or at baseline (since the last assessment)
  * Patients who exhibited suicidal behavior on C-SSRS at screening (for the past 2 years) or at baseline (since the last assessment)
  * Patients who present a serious risk of suicide based on the judgment of the investigator
* Patients presenting tardive dyskinesia at the time of informed consent, as determined by a score of 3 (moderate) or 4 (severe) for Item 8 (severity of abnormal movements) of the AIMS at screening or at baseline
* Patients with a score of 5 (severe akathisia) in the BARS global clinical assessment of akathisia at screening or at baseline
* Patients who meet either of the following criteria between 30 days before screening and the start of screening*

  * Not including the start date of screening

    1. Received 2 or more antipsychotics, each at doses equivalent to ≥ 600 mg/day of chlorpromazine
    2. Received a mean daily dose equivalent to > 800 mg/day**,*** of chlorpromazine

       '**If multiple antipsychotics are taken in the same day, this is to be the combined equivalent dose.

       ***This does not include administration of antipsychotic medication at doses equivalent to less than 100 mg/day of chlorpromazine, which are not expected to have any antipsychotic effect. Chlorpromazine equivalent doses are based on Equivalent Conversion Table for Antipsychotics, as specified separately.
* Patients with a diagnosis of a concurrent mental disorder besides schizophrenia (schizoaffective disorder, major depressive disorder, bipolar I disorder, bipolar II disorder, general anxiety disorder, obsessive-compulsive disorder, post-traumatic stress disorder, dementia or mild neurocognitive disorder, personality disorder, etc) based on DSM-5®. However, this exclusion does not apply to the following:

  • Caffeine- or tobacco-related disorders
* Patients who have met the DSM-5® diagnostic criteria for substance-related or addictive disorder, including alcohol and benzodiazepines but excluding caffeine and tobacco, within 180 days before commencement of investigational medicinal product (IMP) administration
* Patients who have a clinically significant neurological, hepatic, renal, metabolic, hematological, immunological, cardiovascular, pulmonary, or gastrointestinal disorder. Medical conditions that are minor or well-controlled may be considered acceptable if the condition does not interfere with safety and efficacy assessments.
* Patients with known hypersensitivity or intolerance to brexpiprazole or patients with confirmed resistance to brexpiprazole therapy. Patients who have received brexpiprazole to treat the current episode.
* Patients judged by the investigator to be unsuitable for participation in the trial.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 450 (Estimated)
Dates: Start 2022-07-21 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in the Positive and Negative Syndrome Scale (PANSS) total score at last visit of the double-blind period | Baseline and Week 7

CONTACTS AND LOCATIONS:
Overall Officials: Takeshi Tsunoda, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Hayakawa Clinic, Kure-shi, Japan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article Publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com.